CLINICAL TRIAL: NCT05029362
Title: SmokefreeSGM, A Text-based Smoking Cessation Intervention for Sexual and Gender Minority Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Irene Tami-Maury, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-0318 (aim 2); 1K22CA237639 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: LGBTQI
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beta testing group (Other)
  Interventions: Behavioral: SmokefreeSGM

INTERVENTIONS:
Behavioral: SmokefreeSGM — Participants will have access to a text-based smoking cessation program tailored to sexual minority individuals (SmokefreeSGM). The text-based program will be beta-tested by these participants for a period of 2 weeks before and 10 weeks after their quit date. Messages originated from the text-based smoking cessation program will be sent by a fictitious quit coach who will offer evidence-based advice on quitting smoking based on real-life experiences of sexual minority individuals.

SUMMARY:
The purpose of this study is to pretest the design of a text-based smoking cessation program tailored to sexual minority individuals.

ELIGIBILITY:
Inclusion Criteria:

* Smoke five or more cigarettes per day, has smoked at least 100 cigarettes in their lifetime and smokes everyday
* Have an interest in quitting smoking in the next 15 days
* Have a cellphone number with an unlimited short messaging service (SMS) plan
* Have US mailing and email addresses
* Positive cotinine saliva test results

Exclusion Criteria:

* Individuals who are found to have a prepaid cell phone
* Individuals who are found to have a cellphone number that does not work or is registered to someone else
* Pregnant or breastfeeding women
* Contraindication for nicotine patch
* Regular use of tobacco products other than cigarettes
* Current use of tobacco cessation medications
* Enrolled in another smoking cessation study
* Non-English speakers
* Having inadequate equipment/device (webcam, speakers, mic) for participating in telehealth sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as a lesbian, gay, or bisexual individual
Enrollment: 18 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tami-Maury, DMD, MSc, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tami-Maury I, Klaff R, Hussin A, Smith NG, Chang S, McNeill L, Reitzel LR, Shete S, Abroms LC. A Text-Based Smoking Cessation Intervention for Sexual and Gender Minority Groups: Protocol for a Feasibility Trial. JMIR Res Protoc. 2022 Dec 9;11(12):e42553. doi: 10.2196/42553. PMID 36485022

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Beta Testing Group
Started | 18
Completed | 9
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Beta Testing Group
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12.16)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7
  Female | 7
  Nonbinary, genderfluid, or genderqueer | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4
  Non-Hispanic White | 9
  Non-Hispanic Black | 3
  Non-Hispanic Other | 2
Sexual Orientation [Count of Participants; unit: Participants]
  Lesbian/gay woman/Women who have sex with women | 2
  Gay man/Men who have sex with men | 5
  Bisexual female | 5
  Bisexual Male | 3
  Other | 3
Work Status [Count of Participants; unit: Participants]
  Not working | 1
  Working full time | 13
  Working part-time | 4
Education [Count of Participants; unit: Participants]
  Some college or less | 13
  College or higher | 5
Marital status [Count of Participants; unit: Participants]
  Single/separated/divorced/widowed | 17
  married/living with significant other | 1
Children in household [Count of Participants; unit: Participants]
  Yes | 3
  No | 15
Age at which participant first smoked [Mean (Standard Deviation); unit: years] | 14.8 (2.96)
Number of Participants who live with other smokers [Count of Participants; unit: Participants] | 2
Number of times participants tried to quit smoking [Count of Participants; unit: Participants]
  More than 5 times | 8
  Between 1 and 5 times | 9
  Never | 1
Nicotine dependence as assessed by the Fagerstrom Test for Nicotine Dependence [Count of Participants; unit: Participants] — The Fagerström Test for Nicotine Dependence (FTND) is a standard instrument for assessing the intensity of physical addiction to nicotine. The total score ranges from 0 to 10. Participants were categorized as low (less than 4), moderate(between 4 and 6) or high (greater than 6) nicotine dependence based on their FTND score.
  Participants
    high dependence on nicotine | 5
    moderate dependence | 7
    low dependence | 6
Level of Smoking [Count of Participants; unit: Participants]
  Heavy smoker (>10 cigarettes per day) | 7
  Light smoker (less than or equal to 10 cigarettes per day) | 11

OUTCOME MEASURES:

1. Primary Outcome: Perceived Usability as Assessed by the System Usability Scale (SUS)
Description: The 10-item System Usability Scale (SUS) was used to assess the usability of the SmokefreeSGM text messaging program. Total score ranges from 0 to 100, with a higher score indicating greater acceptability and a score above 75 indicating that the program is perceived as acceptable.
Time Frame: 1 month after quit date
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta Testing Group
Number analyzed (Participants) | 9
score on a scale | 81.67 (15.46)

2. Secondary Outcome: Engagement as Assessed by the Number of Text Messages Sent and Received by Study Participants After Enrollment.
Description: A participant's engagement rate was determined by dividing the total number of participant responses to the bidirectional text messages (numerator) by the total number of bidirectional text messages sent by the text-based platform (denominator). Participants who had rates ≤33.3% were classified as having low engagement, 33.3-66.6% moderate engagement, and ≥66.7% high engagement. Data are reported categorically as number of participants who have low, moderate, or high engagement.
Time Frame: 1 month after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Testing Group
Number analyzed (Participants) | 18
Participants
  Low engagement | 5
  moderate engagement | 3
  high engagement | 10

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Beta Testing Group
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT05029362/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT05029362/ICF_002.pdf